CLINICAL TRIAL: NCT03353610
Title: The PSVT Place Registry. Paroxysmal Supraventricular Tachycardia (PSVT) Registry: A Web-based, Prospective, Observational Study.
Brief Title: The PSVT Place Registry.Paroxysmal Supraventricular Tachycardia (PSVT) Registry.
Status: Terminated | Type: Observational
Why Stopped: Termination due to lack of adequate enrollment
Sponsor: Milestone Pharmaceuticals Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: MSP-2017-1141
Record Dates: First submitted 2017-11-13; First posted 2017-11-27 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Paroxysmal Supraventricular Tachycardia (PSVT)
Keywords: Tachycardia; PSVT episodes
MeSH Terms: conditions — Tachycardia, Ventricular; Tachycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient-reported PSVT.: Participants who recorded a PSVT diagnosis.
- Suspected PSVT.: Participants who do not record a PSVT diagnosis.
- Other subgroups.: Subgroups also may be examined ( PSVT-episode characteristics, use of a self-management technique for PSVT at home (on their own) to return heart rate back to normal).The sample size, however, may limit the extent of any subgroup analyses.

SUMMARY:
Paroxysmal supraventricular tachycardia (PSVT) is a sporadic, sudden, and recurring tachycardia that is caused by an altered electrical conductivity in the heart. It causes palpitations and a rapid heart rate, which may induce fear in the patient and negatively impact the patient's quality of life. Therefore, most patients experience not only physical symptoms of PSVT, but also dramatic psychological burdens.

As PSVT drug development efforts advance, it has become increasingly important to document the impact of PSVT in a systematic way, in terms of the disease natural history and clinical characteristics of PSVT episodes, as well as the psychological impact of the condition as reported by patients over time. In order to meet the needs for ongoing, systematic data collection on PSVT, a multinational registry, The PSVT Place Registry (www.PSVTPlaceRegistry.com), is being implemented and will be initially comprised of data entered directly by patients. The long-term registry is designed with a participant-focused approach to enable continuity of data collection and minimization of impact from changes of participants' health care providers. The registry may be expanded at a later time to include physician-reported data.

The information from the registry is planned to be a resource for participants with PSVT, their families and support networks, their doctors, and the research community to better understand PSVT-related symptoms and awareness, PSVT diagnoses, patient self-management, medical treatments for PSVT, and impact of PSVT on quality of life from the patient perspective.

ELIGIBILITY:
Inclusion Criteria:

A participant must meet all of the following criteria to be eligible for participation in the study:

* Adult male or female.
* Participant has suspected PSVT as per the online prescreening assessment.
* Participant lives in a country in which the registry is being conducted.
* Participant has signed the informed consent form indicating he/she is able to complete the online registry data collection forms on his/her own.

Exclusion Criteria:

* Participant does not have an email address.
* Participant does not set up a user account.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult male and females, with suspected PSVT as per online prescreening assessment, who are willing to participate in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Patient Reported Frequency of Recurring PSVT Episodes Using a Patient-Directed Survey Developed by Milestone Pharmaceuticals. | Baseline, then every three months for up to 10 years
  The patient is able to report the frequency (number of PSVT episodes per day, week, month, etc.) for each of their recurring PSVT episodes. Changes in PSVT episode frequency over time will also be assessed.
Patient Reported Duration of Recurring PSVT Episodes Using a Patient-Directed Survey Developed by Milestone Pharmaceuticals. | Baseline, then every three months for up to 10 years.
  The patient is able to report the duration (seconds, minutes, hours, etc.) for each of their recurring PSVT episodes. Changes in PSVT episode duration over time will also be assessed.
Patient Reported Severity of Recurring PSVT Episodes Using a Patient-Directed Survey Developed by Milestone Pharmaceuticals. | Baseline, then every three months for up to 10 years.
  The patient is able to report the severity (1, not severe at all - 5, extremely severe) for each of their recurring PSVT episodes. Changes in PSVT episode severity over time will also be assessed.

SECONDARY OUTCOMES:
Patient Reported Descriptions of the Symptoms to Characterize Their Recurring PSVT Episodes Using a Patient-Directed Survey Developed by Milestone Pharmaceuticals. | Baseline, then every three months for up to 10 years.
  The patient is able to report the most common symptoms that they use to describe each of their recurring PSVT episodes. Changes in PSVT episode symptoms over time will also be assessed.
Patient Reported Descriptions of Health Resource Utilization to Manage Their Recurring PSVT Episodes Using a Patient-Directed Survey Developed by Milestone Pharmaceuticals. | Baseline, then every three months for up to 10 years.
  The patient is able to report physician visits, emergency room visits, hospital admissions, surgical interventions, medication use, monitoring device use, and patient self-management techniques, which are used to assess health resource utilization for each of their recurring PSVT episodes.

OTHER OUTCOMES:
Patient Reported Measures of Mobility, Self-care, Usual Activities, Pain/Discomfort, and Anxiety/Depression Using the EQ-5D-5L Questionnaire (EuroQol) | Baseline, then every three months for up to 10 years.
  The patient is able to report measures of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression at routine intervals. Changes in EQ-5D-5L scores over time will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Wight, Study Director — Milestone Pharma
Locations (1):
- MAPI, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
The details of the processes of producing and reviewing reports, manuscripts, and presentations based on the data from this registry are described in the registry's publication guidelines.
  The Sponsor and/or designee will prepare periodic summaries of descriptive analyses of the data collected in the registry, as required by the appropriate regulatory authority such as disposition data, summary demographic, clinical, or quality of life data. Since enrollment in the registry is from the general population and may be variable, and there is no planned end date for data collection, there is no pre-specified timeline established for preparation of the data summaries. Thus data may be summarized when there is a sufficient length of data for a sufficient amount of participants to constitute a valuable data presentation. In addition, data may be summarized periodically for presentation at professional conferences and sessions, as appropriate.
Time Frame: The Sponsor and/or designee will submit final study results to the appropriate regulatory authorities, no later than 1 year after closure of the registry by the Sponsor.